CLINICAL TRIAL: NCT00280930
Title: A Randomized Feasibility Study of Letrozole in Postmenopausal Women at Increased Risk for Development of Breast Cancer as Evidenced by High Breast Density
Brief Title: Letrozole in Postmenopausal Women at Increased Risk for Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other); Brigham and Women's Hospital (Other); Massachusetts General Hospital (Other)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: 05-183; NCIC CTG MAP.1
Record Dates: First submitted 2006-01-23; First posted 2006-01-24 (Estimated); Last update posted 2007-01-19 (Estimated); Status verified 2007-01

CONDITIONS: Post-Menopausal; Breast Cancer
Keywords: letrozole; breast cancer; menopause
MeSH Terms: conditions — Breast Neoplasms | interventions — Letrozole

INTERVENTIONS:
Drug: Letrozole

SUMMARY:
The purpose of this study to see what happens to breast density in healthy postmenopausal women after treatment with letrozole in one year, compared with treatment with placebo for one year. Other goals of the study include determining if there is a connection between estrogen level and breast density for women in the study and collecting information about the quality of life of those taking part in the study.

DETAILED DESCRIPTION:
* Patients will be randomized into one of two study groups. Group 1 will receive letrozole and Group 2 will receive placebo. This is a double-blind trial so neither the patient or the doctor will know what treatment group they are assigned to.
* If the patient is in Group 1 they will take letrozole tablets orally once a day with food for one year. Patients in Group 2 will take a placebo tablet orally once a day with food for one year.
* Patients in both groups will also be given calcium tablets (500mg) and vitamin D tablets (400IU) once a day for one year.
* After the initial screening visits, the patient will return to the clinic at 3, 6, 9 and 12 months (a total of up to 6 visits in the first year). There will also be two follow-up visits at 18 and 24 months. For the 3, 9 and 18 month visits, telephone contact instead of a clinic visit is allowed.
* The following tests and procedures will be performed during these visits:

evaluation of side effects; routine blood tests(6, 12, and 24 month visits); urine sample (6 and 12 month visits); complete physical exam including breast exam (12 and 24 month visits); mammogram (12 and 24 month visits); bone marrow density x-ray test (12 and 24 month visits); standard x-rays of the lower back and chest (12 month visit); and a questionnaire about how the patient is feeling (12 and 24 month visits).

* The length of participation in this study is for 1 year of study treatment followed by 1 year of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal status defined as: women >55 years of age-no spontaneous menses for at least 12 months; in women < 55 years-no spontaneous menses within the past 12 months and with an FSH level >34.4 IU/I; bilateral oophorectomy
* If subject had prior invasive breast cancer it must have been surgically removed at the time of orginal diagnosis with no evidence of metastases and the primary tumor may be receptive negative, positive or equivocal
* Baseline mammogram (within 6 months) indicating mammographic density occupying >25% (grade 4/5, 5/6 or 6/6) of the breast tissue
* Baseline breast examination demonstrating no clinical evidence of breast cancer
* Acceptable quality DEXA of the L2-L4 postero-anterior (PA) spine and hup must be performed 6 months of randomization
* Subject is willing and able to complete the quality of life questionnaire in either English or French

Exclusion Criteria:

* Mammogram suspicious for breast cancer (unless subsequently ruled out)
* Patient's with prior malignancies are eligible unless they have metastatic disease
* Uncontrolled metabolic or endocrine disease, cardiovascular disease or malabsorption syndrome
* Current chemotherapy or immunotherapy
* Hormone replacement therapy or Evista (raloxifene) discontinued less than three months before baseline mammogram
* Tamoxifen therapy discontinued less than six months prior to randomization

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2005-10

PRIMARY OUTCOMES:
To determine the proportion of women with breast density of > grade 4 who have a decrease in breast density of at least one grade after treatment with letrozole for one year.

SECONDARY OUTCOMES:
To determine if the decrease in breast density grade is sustained one year after cessation of therapy
to determine if there is a correlation between plasma estrogen profile and breast density at baseline
to determine the percentage of subjects with breast tissue hyperplasia and atypical hyperplasia before and after therapy
to assess change in estrogen profile from baseline and at 1 year and 1 year after cessation of therapy
to assess the general safety of the utilization of letrozole in healthy post-menopausal women for one year
to compare the effects on menopause-specific quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Goss, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts